CLINICAL TRIAL: NCT05365360
Title: Effect of Increasing Fluence on Efficacy of Low Level Laser Therapy for Androgenetic Alopecia, a Randomized Control Trial
Brief Title: Sham LaserCap vs. LaserCap SD vs. LaserCap HD+
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Transdermal Cap, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LLLT Fluence RCT
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Sham LaserCap (Sham Comparator): Sham device
  Interventions: Device: Sham LaserCap
- Lasercap SD (Experimental): Low fluence LLLT
  Interventions: Device: LaserCap SD
- Lasercap HD+ (Experimental): High fluence LLLT
  Interventions: Device: LaserCap HD+

INTERVENTIONS:
Device: LaserCap SD — LaserCap SD
  Arms: Lasercap SD
Device: Sham LaserCap — Sham LaserCap
  Arms: Sham LaserCap
Device: LaserCap HD+ — LaserCap HD+
  Arms: Lasercap HD+

SUMMARY:
Androgenetic alopecia (AGA) is a prevalent disease, occurring in 80% of Caucasian men and 50% of Caucasian women by age 701. Treatments for AGA are limited, and presently the only FDA-approved medications for AGA are topical minoxidil and oral finasteride1.

In addition to medical therapies, FDA-cleared medical devices are now utilized for the treatment of AGA as of 20072. These devices, termed low level laser therapy (LLLT), come in multiple forms including combs, helmets and sports cap wearable devices2. These home-use, wearable devices utilize the ~650 nm wavelength laser light to stimulate the hair follicle mitochondria and thereby promote hair growth, a process termed "photobiomodulation"3.

Recent meta-analyses investigating photobiomodulation and LLLT for AGA have noted an increase in fluence or energy delivered per cm is associated with increased hair density3. However, randomized control trials (RCT) with direct comparison of LLLT devices of different fluences has yet to be performed. Accordingly, in the present study we aim to investigate if increasing fluence in LLLT devices is associated with increased hair density by comparing sham LaserCap to LaserCap SD (1.15 J/cm2, low fluence) and LaserCap HD+ (3.93 J/cm2, high fluence) in RCT.

ELIGIBILITY:
Inclusion criteria:

* 25 years and older
* Men and women with AGA, untreated or with 6-month washout of previous treatments
* Men: Norwood stage IIa - V
* Women: Ludwig I-1 - II-2, or frontal pattern
* All patients: Fitzpatrick skin types I to IV

Exclusion criteria:

* Men: Norwood stage Va, VI, VII
* Women: Ludwig stage III, advanced
* All patients: Fitzpatrick skin types V, VI
* Current use or within the past six month of other treatment for AGA, including topical and oral minoxidil, topical and oral finasteride and dutasteride
* Age 0-25 years

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Target area total hair count at 26 weeks via phototrichogram | 26 weeks

SECONDARY OUTCOMES:
Target area vellus hair count at 26 weeks via phototrichogram | 26 weeks
Target area terminal hair count at 26 weeks via phototrichogram | 26 weeks
Physician assessed improvement via global photography at 26 weeks | 26 weeks
Hair growth rate at 26 weeks via phototrichogram | 26 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Banner University Dermatology, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No